CLINICAL TRIAL: NCT00538525
Title: Phase II Study of Neoadjuvant Chemotherapy With Doxorubicin Followed by Docetaxel-Cisplatin in Locally Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2011-022
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Docetaxel; Cisplatin

ARMS (1):
- Arm 1 (Active Comparator): Doxorubicin, Docetaxel, Cisplatin
  Interventions: Drug: Doxorubicin, Docetaxel, Cisplatin

INTERVENTIONS:
Drug: Doxorubicin, Docetaxel, Cisplatin — Doxorubicin, Docetaxel, Cisplatin

SUMMARY:
Phase II study of neoadjuvant chemotherapy with Doxorubicin followed by Docetaxel-Cisplatin in locally advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced breast cancer

Exclusion Criteria:

* Patients with metastatic breast cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness | overall

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Ezzat, MD, Principal Investigator — KFSH&RC, Riyadh, Saudi Arabia